CLINICAL TRIAL: NCT00934843
Title: Preoperative Corticosteroid Therapy in Neonates Undergoing Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR 17030
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Results first posted 2011-12-09 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-09

CONDITIONS: Congenital Heart Disease; Disorder of Fetus or Newborn
Keywords: Cardiopulmonary Bypass (CPB); System Inflammatory Response; Low Cardiac Output Syndrome (LCOS) in Neonates; Methylprednisolone; Cardiopulmonary Bypass (CPB) in Neonates; Glucocorticoid Use in Neonatal Cardiac Surgery; Steroid
MeSH Terms: conditions — Heart Defects, Congenital; Fetal Diseases; Cardiac Output, Low | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Steroids; Glucocorticoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dose steroid (Experimental): Neonates with congenital heart disease requiring surgery utilizing a cardiopulmonary bypass (CPB) machine in the first month of life that receive ONE dose intravenous methylprednisolone (IVMP) prior to heart surgery.
  Interventions: Drug: methylprednisolone (IVMP)
- Two Dose steroid (Experimental): Neonates with congenital heart disease requiring surgery utilizing a cardiopulmonary bypass (CPB) machine in the first month of life that receive TWO doses intravenous methylprednisolone (IVMP) prior to heart surgery.Compare the effects and preoperative and intraoperative IVMP to intraoperative IVMP alone on the inflammatory response to CPB cardiopulmonary bypass. The hypothesis is that neonates treated with preoperative IVMP as well as the standard intraoperative IVMP will have decreased production of pro-inflammatory cytokines.
  Interventions: Drug: methylprednisolone (two doses IVMP)

INTERVENTIONS:
Drug: methylprednisolone (IVMP) — Neonates with congenital heart disease requiring surgery utilizing a cardiopulmonary bypass (CPB)machine in the first month of life that receive ONE doses intravenous methylprednisolone (IVMP) prior to heart surgery.Compare the effects and preoperative and intraoperative IVMP (2 dose steroid)to intraoperative IVMP alone (single dose steroid) on the inflammatory response to CPB cardiopulmonary bypass.
  Other Names: Solumedrol; Steroid; glucocorticoid
  Arms: Single dose steroid
Drug: methylprednisolone (two doses IVMP) — Neonates with congenital heart disease requiring surgery utilizing a cardiopulmonary bypass (CPB)machine in the first month of life that receive TWO doses intravenous methylprednisolone (IVMP) prior to heart surgery.Compare the effects and preoperative and intraoperative IVMP to intraoperative IVMP alone on the inflammatory response to CPB cardiopulmonary bypass. The hypothesis is that neonates treated with preoperative IVMP as well as the standard intraoperative IVMP will have decreased production of pro-inflammatory cytokines.
  Other Names: Solumedrol; Steroid; glucocorticoid
  Arms: Two Dose steroid

SUMMARY:
Randomized controlled trial of the use of glucocorticoids to improve the clinical course of neonates post-cardiopulmonary bypass (CPB).

DETAILED DESCRIPTION:
This study proposes a randomized controlled trial of the use of glucocorticoids to improve the clinical course of neonates post-cardiopulmonary bypass (CPB). The study will focus on neonates for a few reasons. Although their post-CPB clinical course is typically more severe and intensive care unit (ICU) care more prolonged than older children, their modes of morbidity are also well characterized. Further, the high level of severity itself provides a substrate for identifying the positive effects of a particular therapy. Finally, a therapy identified as beneficial has the greatest potential for benefit in this vulnerable population. The well characterized scenario of low cardiac output syndrome (LCOS) will be used as the primary endpoint, while a variety of secondary endpoints will be related to the biochemical anti-inflammatory effects of therapy, ICU care and late neurological outcome.

ELIGIBILITY:
Inclusion Criteria:

* Neonates Age </= 1 month
* Scheduled to undergo cardiac surgery involving Cardiopulmonary Bypass (CPB) (reparative or palliative procedures)
* Inpatient Status at MUSC a minimum of 8 hours prior to planned surgery

Exclusion Criteria:

* Prematurity: </= 36 weeks post gestational age at time of surgery
* Treatment with steroids, other than inhaled forms, in the two weeks prior to scheduled surgery
* Participation in research studies involving the evaluation of investigational drugs within 30 days of randomization
* Suspected infection that would contraindicate steroid use (eg - Herpes)
* Known hypersensitivity to IVMP or one of its components or other contraindication to steroid therapy (e.g., gastrointestinal bleeding)
* Preoperative use of mechanical circulatory support or active resuscitation at the time of proposed randomization
* Inability to begin the pre-operative study drug at least 8 hours prior to surgery

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2007-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Graham, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Hoffman TM, Wernovsky G, Atz AM, Kulik TJ, Nelson DP, Chang AC, Bailey JM, Akbary A, Kocsis JF, Kaczmarek R, Spray TL, Wessel DL. Efficacy and safety of milrinone in preventing low cardiac output syndrome in infants and children after corrective surgery for congenital heart disease. Circulation. 2003 Feb 25;107(7):996-1002. doi: 10.1161/01.cir.0000051365.81920.28. PMID 12600913
- [Background] Thompson LD, McElhinney DB, Findlay P, Miller-Hance W, Chen MJ, Minami M, Petrossian E, Parry AJ, Reddy VM, Hanley FL. A prospective randomized study comparing volume-standardized modified and conventional ultrafiltration in pediatric cardiac surgery. J Thorac Cardiovasc Surg. 2001 Aug;122(2):220-8. doi: 10.1067/mtc.2001.114937. PMID 11479493
- [Background] Turley K, Mavroudis C, Ebert PA. Repair of congenital cardiac lesions during the first week of life. Circulation. 1982 Aug;66(2 Pt 2):I214-9. PMID 7083544
- [Background] Frantz S, Bauersachs J, Kelly RA. Innate immunity and the heart. Curr Pharm Des. 2005;11(10):1279-90. doi: 10.2174/1381612053507512. PMID 15853684
- [Background] Chaney MA. Corticosteroids and cardiopulmonary bypass : a review of clinical investigations. Chest. 2002 Mar;121(3):921-31. doi: 10.1378/chest.121.3.921. PMID 11888978
- [Background] Checchia PA, Bronicki RA, Costello JM, Nelson DP. Steroid use before pediatric cardiac operations using cardiopulmonary bypass: an international survey of 36 centers. Pediatr Crit Care Med. 2005 Jul;6(4):441-4. doi: 10.1097/01.PCC.0000163678.20704.C5. PMID 15982431
- [Background] Dickerson HA, Chang AC. Steroids and low cardiac output syndrome after cardiac surgery in children. Pediatr Crit Care Med. 2005 Jul;6(4):495-6. doi: 10.1097/01.pcc.0000164640.09454.61. No abstract available. PMID 16003215
- [Background] Mann DL. Targeted anticytokine therapy and the failing heart. Am J Cardiol. 2005 Jun 6;95(11A):9C-16C; discussion 38C-40C. doi: 10.1016/j.amjcard.2005.03.007. PMID 15925559
- [Background] Tuckermann JP, Kleiman A, McPherson KG, Reichardt HM. Molecular mechanisms of glucocorticoids in the control of inflammation and lymphocyte apoptosis. Crit Rev Clin Lab Sci. 2005;42(1):71-104. doi: 10.1080/10408360590888983. PMID 15697171
- [Background] Checchia PA, Backer CL, Bronicki RA, Baden HP, Crawford SE, Green TP, Mavroudis C. Dexamethasone reduces postoperative troponin levels in children undergoing cardiopulmonary bypass. Crit Care Med. 2003 Jun;31(6):1742-5. doi: 10.1097/01.CCM.0000063443.32874.60. PMID 12794414
- [Background] Schroeder VA, Pearl JM, Schwartz SM, Shanley TP, Manning PB, Nelson DP. Combined steroid treatment for congenital heart surgery improves oxygen delivery and reduces postbypass inflammatory mediator expression. Circulation. 2003 Jun 10;107(22):2823-8. doi: 10.1161/01.CIR.0000070955.55636.25. Epub 2003 May 19. PMID 12756159
- [Background] Varan B, Tokel K, Mercan S, Donmez A, Aslamaci S. Systemic inflammatory response related to cardiopulmonary bypass and its modification by methyl prednisolone: high dose versus low dose. Pediatr Cardiol. 2002 Jul-Aug;23(4):437-41. doi: 10.1007/s00246-002-0118-3. PMID 12170362
- [Background] Mott AR, Fraser CD Jr, Kusnoor AV, Giesecke NM, Reul GJ Jr, Drescher KL, Watrin CH, Smith EO, Feltes TF. The effect of short-term prophylactic methylprednisolone on the incidence and severity of postpericardiotomy syndrome in children undergoing cardiac surgery with cardiopulmonary bypass. J Am Coll Cardiol. 2001 May;37(6):1700-6. doi: 10.1016/s0735-1097(01)01223-2. PMID 11345387
- [Background] Bronicki RA, Backer CL, Baden HP, Mavroudis C, Crawford SE, Green TP. Dexamethasone reduces the inflammatory response to cardiopulmonary bypass in children. Ann Thorac Surg. 2000 May;69(5):1490-5. doi: 10.1016/s0003-4975(00)01082-1. PMID 10881828
- [Background] Lindberg L, Forsell C, Jogi P, Olsson AK. Effects of dexamethasone on clinical course, C-reactive protein, S100B protein and von Willebrand factor antigen after paediatric cardiac surgery. Br J Anaesth. 2003 Jun;90(6):728-32. doi: 10.1093/bja/aeg125. PMID 12765886
- [Background] Ungerleider R. Practice patterns in neonatal cardiopulmonary bypass. Semin Thorac Cardiovasc Surg Pediatr Card Surg Annu. 2004;7:172-9. doi: 10.1053/j.pcsu.2004.02.022. PMID 15283366
- [Background] Parr GV, Blackstone EH, Kirklin JW. Cardiac performance and mortality early after intracardiac surgery in infants and young children. Circulation. 1975 May;51(5):867-74. doi: 10.1161/01.cir.51.5.867. PMID 235375
- [Background] Wernovsky G, Wypij D, Jonas RA, Mayer JE Jr, Hanley FL, Hickey PR, Walsh AZ, Chang AC, Castaneda AR, Newburger JW, Wessel DL. Postoperative course and hemodynamic profile after the arterial switch operation in neonates and infants. A comparison of low-flow cardiopulmonary bypass and circulatory arrest. Circulation. 1995 Oct 15;92(8):2226-35. doi: 10.1161/01.cir.92.8.2226. PMID 7554206
- [Background] Friedman WF. Congenital heart disease in infancy and childhood. Heart Disease - A Textbook of Cardiovascular Medicine. 4th ed. Philadelphia, PA. W.B. Saunders Co.; 1992. p. 894.
- [Background] Greeley WJ, Kern FH, Ungerleider RM, Boyd JL 3rd, Quill T, Smith LR, Baldwin B, Reves JG. The effect of hypothermic cardiopulmonary bypass and total circulatory arrest on cerebral metabolism in neonates, infants, and children. J Thorac Cardiovasc Surg. 1991 May;101(5):783-94. PMID 2023435
- [Background] Kulik TJ, Moler FW, Palmisano JM, Custer JR, Mosca RS, Bove EL, Bartlett RH. Outcome-associated factors in pediatric patients treated with extracorporeal membrane oxygenator after cardiac surgery. Circulation. 1996 Nov 1;94(9 Suppl):II63-8. PMID 8901721
- [Derived] Schroeder LW, Buckley JR, Stroud RE, Martin RH, Nadeau EK, Barrs R, Graham EM. Plasma Neutrophil Gelatinase-Associated Lipocalin Is Associated With Acute Kidney Injury and Clinical Outcomes in Neonates Undergoing Cardiopulmonary Bypass. Pediatr Crit Care Med. 2019 Oct;20(10):957-962. doi: 10.1097/PCC.0000000000002035. PMID 31206501
- [Derived] Graham EM, Atz AM, McHugh KE, Butts RJ, Baker NL, Stroud RE, Reeves ST, Bradley SM, McGowan FX Jr, Spinale FG. Preoperative steroid treatment does not improve markers of inflammation after cardiac surgery in neonates: results from a randomized trial. J Thorac Cardiovasc Surg. 2014 Mar;147(3):902-8. doi: 10.1016/j.jtcvs.2013.06.010. Epub 2013 Jul 16. PMID 23870160
- [Derived] Butts RJ, Scheurer MA, Zyblewski SC, Wahlquist AE, Nietert PJ, Bradley SM, Atz AM, Graham EM. A composite outcome for neonatal cardiac surgery research. J Thorac Cardiovasc Surg. 2014 Jan;147(1):428-33. doi: 10.1016/j.jtcvs.2013.03.013. Epub 2013 Apr 12. PMID 23587468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All inpatient neonates (≤ 30 days of age), scheduled to undergo cardiac surgery involving cardiopulmonary bypass from the time period of July 2007 through July 2009 were eligible for this study.
Groups:
- MP Single Dose: Neonates with congenital heart disease requiring surgery utilizing a cardiopulmonary bypass (CPB) machine in the first month of life that receive ONE dose (operatively)intravenous methylprednisolone (IVMP, 30 mg/kg) prior to heart surgery.
- MP Two Dose: Neonates with congenital heart disease requiring surgery utilizing a cardiopulmonary bypass (CPB) machine in the first month of life that receive TWO (8 hours preoperatively and operatively) doses intravenous methylprednisolone (IVMP, 30 mg/kg/dose) prior to heart surgery.
Period: Overall Study
Arm/Group | MP Single Dose | MP Two Dose
Started | 37 | 40
Completed | 37 | 39 (1 subject discontinued intervention, surgery plan changed and did not require CPB)
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MP Single Dose | MP Two Dose | Total
Number analyzed (Participants) | 37 | 40 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37 | 40 | 77
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: days] | 8.2 (5.0) | 9.4 (6.3) | 8.8 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 19 | 21 | 40
Region of Enrollment [Number; unit: participants]
  United States | 37 | 40 | 77

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint: Number of Participants With Low Cardiac Output Syndrome (LCOS) or Death at 36 Hours From Admission to the Intensive Care Unit (ICU) After Surgery.
Description: The presence of low cardiac output syndrome (LCOS) was defined by the same definition used in the PRIMACORP study (Hoffman TM.et.al. Circulation 2003 107:996-1002). Specifically, if there were clinical signs and symptoms of low cardiac output (e.g., tachycardia, oliguria, cold extremities, cardiac arrest, etc.) which required one or more of the following interventions: mechanical circulatory support, the escalation of existing pharmacological circulatory support to >100% over baseline, or the initiation of new pharmacological circulatory support.
Time Frame: 36 hours
Measure: Number; unit: participants
Groups:
- MP Single Dose: Neonates scheduled for cardiac surgery that were randomly assigned to receive Single Dose (operatively) methylprednisolone (30 mg/kg/dose)
- MP Two Dose: Neonates scheduled for cardiac surgery that were randomly assigned to receive Two Dose (8 hours preoperatively and operatively) methylprednisolone (30 mg/kg/dose).
Arm/Group | MP Single Dose | MP Two Dose
Number analyzed (Participants) | 37 | 39
participants | 17 | 15
Statistical Analysis 1: Comparison: MP Single Dose vs MP Two Dose; The current study was designed with an anticipated enrollment of 87 patients per treatment arm to achieve a statistical power of 80% (1- β) while controlling type I error at 0.05 (α) using a more conservative estimate of LCOS rate in the Single Dose MP group of 33%, and an incidence of LCOS in the Two Dose MP group of 15%; Test type: Superiority or Other; p = 0.35, Multivariate risk computation; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.45 to 1.33]

2. Secondary Outcome: Inotropic Score
Description: The inotropic score was calculated by the equation using drug dosages in micrograms/kg/min, (dopamine+dobutamine) + (milrinonex10) + (epinephrinex100) and recorded hourly upon arrival to the ICUthrough 36 hours postoperatively. The highest score during this timeframe was recorded. This score converts dosages of commonly used inotropic medications into a score. The higher the score the more inotropic medications required. The minimum score would be zero indicating no inotropic medications were used. There is no maximum score.
Time Frame: over the first 36 hours after surgery
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MP Single Dose | MP Two Dose
Number analyzed (Participants) | 37 | 39
Scores on a scale | 14.4 (3.6) | 15.0 (3.9)
Statistical Analysis 1: Comparison: MP Single Dose vs MP Two Dose; Test type: Superiority or Other; p = 0.43, ANCOVA — A repeated measures analysis of variance framework was used for longitudinal analysis of inotrope score. In order to identify potential confounding variables, a variable was considered a relevant covariate and added into the model with a p ≤ 0.15

3. Secondary Outcome: Number of Participants Who Died Between 36 Hours and 30 Days Following Cardiac Surgery
Description: Number of participants who died of any cause between 36 hours and 30 days following cardiac surgery
Time Frame: at 36 hours and 30 days
Measure: Number; unit: participants
Arm/Group | MP Single Dose | MP Two Dose
Number analyzed (Participants) | 37 | 39
participants | 1 | 0

4. Secondary Outcome: Urine Output
Description: Total urine output in mL over the first 36 hours after cardiac surgery
Time Frame: over 36 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MP Single Dose | MP Two Dose
Number analyzed (Participants) | 37 | 39
mL | 498 (227) | 453 (213)
Statistical Analysis 1: Comparison: MP Single Dose vs MP Two Dose; Test type: Superiority or Other; p = 0.052, ANCOVA — Analysis of variance/covariance models were used to test both unadjusted and multivariable relationships between treatment groups for diuresis

5. Secondary Outcome: Total Intake/Output of Fluid
Description: Total amount of all fluids in and out during the first 36 hours postoperatively in mL.
Time Frame: over 36 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MP Single Dose | MP Two Dose
Number analyzed (Participants) | 37 | 39
mL
  Total Fluid in at 36 hr | 575 (145) | 586 (156)
  Total Fluid out at 36 hr | 600 (250) | 558 (203)
Statistical Analysis 1: Comparison: MP Single Dose vs MP Two Dose; Test type: Superiority or Other; p = 0.047, ANCOVA; Analysis of variance/covariance models were used to test both unadjusted and multivariable relationships between treatment groups for diuresis

ADVERSE EVENTS:
Arm/Group | MP Single Dose | MP Two Dose
Serious Adverse Events (participants affected / at risk) | 1/37 | 0/39
Other Adverse Events (participants affected / at risk) | 6/37 | 10/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MP Single Dose (N=37) | MP Two Dose (N=39)
Death (Cardiac disorders) | 1 (1) | 0 (0) — Death within 30 days of operation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MP Single Dose (N=37) | MP Two Dose (N=39)
Infection (Infections and infestations) | 5 (5) | 5 (5) — Documented postoperative culture positive infection
Poor wound healing (Cardiac disorders) | 1 (1) | 5 (5) — Document poor wound healing within 30 days of surgery

LIMITATIONS AND CAVEATS:
Limitations of the current study include the lack of a true placebo group. Thus recommendations for or against intraoperative MP can not be made. The results of our trial do not preclude the efficacy of other glucocorticoid regimens.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes